CLINICAL TRIAL: NCT02458300
Title: FIBARRIX "Clinical Evaluation of the Response to Chest Physiotherapy in Infants With Acute Bronchiolitis"
Brief Title: Clinical Evaluation of the Response to Chest Physiotherapy in Children With Acute Bronchiolitis
Acronym: FIBARRIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Enrique Conesa Segura, PT, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIBARRIX
Record Dates: First submitted 2015-05-20; First posted 2015-06-01 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2015-05

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; Chest; Physical therapy
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (Placebo Comparator): Nebulized hypertonic saline. Aspiration of secretions
  Interventions: Other: Nebulization of hypertonic saline; Other: Aspiration of secretions
- Intervention Arm. (Active Comparator): Nebulization of hypertonic saline. Application of Prolonged slow expiration technique (PSE) expiratory volume. Patient coughing Provocation (TP) Inspiratory maneuver to rhinopharyngeal cleaning DRR Aspiration of secretions
  Interventions: Other: Nebulization of hypertonic saline; Other: Prolonged slow expiration technique (PSE); Other: Patient coughing Provocation (TP); Other: inspiratory maneuver to rhinopharyngeal cleaning DRR; Other: Aspiration of secretions

INTERVENTIONS:
Other: Nebulization of hypertonic saline — application of hypertonic saline serum through a mask fogging or a box fogging
Other: Prolonged slow expiration technique (PSE) — Passive expiratory aid implemented baby. the child is placed supine on a hard surface. Thoracoabdominal slow manual pressure that begins at the end of a spontaneous and continuous exhalation to residual volume is exercised. Oppose reaches 2 or 3 breaths. Vibrations can accompany the art. The goal is to achieve a greater expiratory volume.
  Arms: Intervention Arm.
Other: Patient coughing Provocation (TP) — Tp is based on the mechanism reflects cough induced by stimulation of the buttons on the wall of the trachea extrathoracic mechanoreceptors. The child is placed supine. A short pressure is done with the thumb on the tracheal conduit (in the sternal notch) at the end of inspiration, or at the beginning of expiration. With the other hand holding the abdominal region we prevent the dissipation of energy and make the explosion tussive more effective. It is done after the PSE.
  Arms: Intervention Arm.
Other: inspiratory maneuver to rhinopharyngeal cleaning DRR — After the inspiratory reflection following the PSE, the TP or crying. At the end of expiratory time the child's mouth is closed with the back of his hand just finished his chest support, raising the jaw and forcing the child to an inspiration with the nose
  Arms: Intervention Arm.
Other: Aspiration of secretions — Suctioning with a probe by a vacuum system installed on the wall.

SUMMARY:
The objective of this study is to evaluate the clinical response of children diagnosed with acute bronchiolitis, relative to a chest physiotherapy protocol. Comparing this treatment with standard care of the nursing staff and auxiliaries of infants patients aged 1 month to 2 years.

DETAILED DESCRIPTION:
This randomized clinical trial has an intervention group and a control group. All treatment will be made by physiotherapist with extensive clinical experience and training in techniques of Chest physiotherapy (CPT). Performing at least one session per day during the time of patient admission. This session takes an average of about 15 minutes, begins by fogging of hypertonic saline, and ends with the nasal and oral suction of the patient. The evaluation of clinical data is done 10 minutes before, 10 minutes later, 2 hours after physiotherapy treatment. The evaluation will be do it for a doctor who will, in all patients, a clinical examination that includes all items scale clinical severity of acute bronchiolitis.

Patient Registries:

SELECTION OF THE POPULATION Reference population. Patients diagnosed acute viral bronchiolitis during the conduct of the trial and have been admitted to the University Hospital Virgin of Arrixaca.

Sample size

The sample calculation was done considering a reduction of 2 points after physiotherapy in bronchiolitis severity scale. Whereas:

Variances: sames Detect mean difference: 2,000 Common standard deviation: 2,370 Ratio of sample sizes: 1,00 Confidence level: 95,0%

The standard deviation values were obtained from: JM Fernández Ramos et al Validation of a clinical scale of severity of acute bronchiolitis. An Pediatr (Barc). 2014; 81 (1): 3-8, article in which the mean and standard deviation (SD) score of patients admitted was 7 ± 2.37. There are no items to compare this scale before and after treatment, so the investigators have assumed that value of common standard deviation (SD) and whereas a decrease of 2 points on the scale post-physical therapy would be clinically relevant.

Power (%) Sample size Cases Control Total 85,0 27 27 54 90 31 31 62

Finally it was decided to increase to 60 cases / group considering that the number of losses may be higher (the investigators calculate 50%).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the pediatric intensive care unit or pediatric nursing unit. Which they are diagnostic of acute viral bronchiolitis (AVB).

Exclusion Criteria:

* Presence of cyanotic congenital heart disease no longer for comparing the constants.
* Relative or absolute contraindication CPT techniques included in the protocol.

  * Patients diagnosed with moderate or severe gastroesophageal reflux since the PSE gastroesophageal reflux can accentuate a previously exist.
  * Patients with laryngeal diseases caused because the cough is a technique that is applied directly to the tracheal wall and can affect the larynx.
  * Absence of cough reflects and presence of laryngeal stridor is a contraindication to chest physiotherapy in general.
  * Systematic presence of gag reflex as the aspiration of secretions and coughing caused nasobucales stimulate this reflex

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of a physiotherapy treatment with clinical severity scale of a patient diagnosed with acute viral bronchiolitis | Participants will be followed for the duration of hospital stay, an expected average of 7 days

SECONDARY OUTCOMES:
Assess the variation of score, a scale of severity of acute viral bronchiolitis, after intervention protocols | Participants will be followed for the duration of hospital stay, an expected average of 7 days
Analyze a inquiry of subjective opinion, completed by parents or tutors at the end of treatment | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  A questionnaire was filled out by parents or guardians of patients. After, the results of the survey will be analyzed by means of SPSS software
To quantify the changes in clinical score severity scale. | Participants will be followed for the duration of hospital stay, an expected average of 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Enrique E Conesa Segura, PT, Principal Investigator — MurciaSalud; Susana Beatriz S Reyes Dominguez, PhD,MD, Principal Investigator — MurciaSalud; José J Rios Diaz, PhD, BiolSc, PT, Study Chair — Universidad Católica San Antonio de Murcia; Eduardo E Ramos Elbal, MD, Study Chair — MurciaSalud; Cristina C Palazón Carpe, MD, Study Chair — MurciaSalud; Maria Ángeles M Ruiz Pacheco, MD, Study Chair — MurciaSalud; Jaume J Enjuanes Llovet, MD, Study Chair — MurciaSalud; Sara S Francés Tarazona, MD, Study Chair — MurciaSalud; Sebastián S Gil Garcia, PT, Study Chair — MurciaSalud; Maía de los Ángeles M Martinez-Salazar Arboleas, PT, Study Chair — MurciaSalud

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aherne W, Bird T, Court SD, Gardner PS, McQuillin J. Pathological changes in virus infections of the lower respiratory tract in children. J Clin Pathol. 1970 Feb;23(1):7-18. doi: 10.1136/jcp.23.1.7. PMID 4909103
- [Background] Bohe L, Ferrero ME, Cuestas E, Polliotto L, Genoff M. [Indications of conventional chest physiotherapy in acute bronchiolitis]. Medicina (B Aires). 2004;64(3):198-200. Spanish. PMID 15239532
- [Background] Fischer GB, Teper A, Colom AJ. Acute viral bronchiolitis and its sequelae in developing countries. Paediatr Respir Rev. 2002 Dec;3(4):298-302. doi: 10.1016/s1526-0542(02)00268-3. PMID 12457599
- [Background] Gajdos V, Katsahian S, Beydon N, Abadie V, de Pontual L, Larrar S, Epaud R, Chevallier B, Bailleux S, Mollet-Boudjemline A, Bouyer J, Chevret S, Labrune P. Effectiveness of chest physiotherapy in infants hospitalized with acute bronchiolitis: a multicenter, randomized, controlled trial. PLoS Med. 2010 Sep 28;7(9):e1000345. doi: 10.1371/journal.pmed.1000345. PMID 20927359
- [Background] Gomes EL, Postiaux G, Medeiros DR, Monteiro KK, Sampaio LM, Costa D. Chest physical therapy is effective in reducing the clinical score in bronchiolitis: randomized controlled trial. Rev Bras Fisioter. 2012 Jun;16(3):241-7. doi: 10.1590/s1413-35552012005000018. Epub 2012 Apr 12. PMID 22499404
- [Background] Hess DR. Airway clearance: physiology, pharmacology, techniques, and practice. Respir Care. 2007 Oct;52(10):1392-6. PMID 17894906
- [Background] Krause MF, Hoehn T. Chest physiotherapy in mechanically ventilated children: a review. Crit Care Med. 2000 May;28(5):1648-51. doi: 10.1097/00003246-200005000-00067. PMID 10834729
- [Background] Lanza FC, Wandalsen G, Dela Bianca AC, Cruz CL, Postiaux G, Sole D. Prolonged slow expiration technique in infants: effects on tidal volume, peak expiratory flow, and expiratory reserve volume. Respir Care. 2011 Dec;56(12):1930-5. doi: 10.4187/respcare.01067. Epub 2011 Jun 17. PMID 21682953
- [Background] McConnochie KM. Bronchiolitis. What's in the name? Am J Dis Child. 1983 Jan;137(1):11-3. No abstract available. PMID 6847951
- [Background] Mellins RB. Pulmonary physiotherapy in the pediatric age group. Am Rev Respir Dis. 1974 Dec;110(6 Pt 2):137-42. doi: 10.1164/arrd.1974.110.6P2.137. No abstract available. PMID 4613219
- [Background] Oberwaldner B. Physiotherapy for airway clearance in paediatrics. Eur Respir J. 2000 Jan;15(1):196-204. doi: 10.1183/09031936.00.15119600. PMID 10678646
- [Background] Postiaux G, Louis J, Labasse HC, Gerroldt J, Kotik AC, Lemuhot A, Patte C. Evaluation of an alternative chest physiotherapy method in infants with respiratory syncytial virus bronchiolitis. Respir Care. 2011 Jul;56(7):989-94. doi: 10.4187/respcare.00721. Epub 2011 Feb 22. PMID 21352671
- [Background] Postiaux G. [Bronchiolitis in infants. What are the techniques of bronchial and upper airway respiratory therapy adapted to infants?]. Arch Pediatr. 2001 Jan;8 Suppl 1:117S-125S. doi: 10.1016/s0929-693x(01)80170-6. No abstract available. French. PMID 11232428
- [Background] Roque i Figuls M, Gine-Garriga M, Granados Rugeles C, Perrotta C. Chest physiotherapy for acute bronchiolitis in paediatric patients between 0 and 24 months old. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD004873. doi: 10.1002/14651858.CD004873.pub4. PMID 22336805
- [Background] Schechter MS. Airway clearance applications in infants and children. Respir Care. 2007 Oct;52(10):1382-90; discussion 1390-1. PMID 17894905
- [Background] van der Schans CP. Forced expiratory manoeuvres to increase transport of bronchial mucus: a mechanistic approach. Monaldi Arch Chest Dis. 1997 Aug;52(4):367-70. PMID 9401368
- [Background] Webb MS, Martin JA, Cartlidge PH, Ng YK, Wright NA. Chest physiotherapy in acute bronchiolitis. Arch Dis Child. 1985 Nov;60(11):1078-9. doi: 10.1136/adc.60.11.1078. PMID 3907510
- [Background] Wohl ME, Chernick V. State of the art: bronchiolitis. Am Rev Respir Dis. 1978 Oct;118(4):759-81. doi: 10.1164/arrd.1978.118.4.759. No abstract available. PMID 212970
- [Background] Zach MS, Oberwaldner B. Chest physiotherapy--the mechanical approach to antiinfective therapy in cystic fibrosis. Infection. 1987;15(5):381-4. doi: 10.1007/BF01647750. PMID 3319913
- [Derived] Roque-Figuls M, Gine-Garriga M, Granados Rugeles C, Perrotta C, Vilaro J. Chest physiotherapy for acute bronchiolitis in paediatric patients between 0 and 24 months old. Cochrane Database Syst Rev. 2023 Apr 3;4(4):CD004873. doi: 10.1002/14651858.CD004873.pub6. PMID 37010196